CLINICAL TRIAL: NCT04124575
Title: Prevalence of Sarcopenia in Patients Admitted to a Swiss University Department of Geriatric Medicine
Brief Title: Prevalence of Sarcopenia in Geriatric Patients
Status: Completed | Type: Observational
Sponsor: University Department of Geriatric Medicine FELIX PLATTER (Other)
Responsible Party: Sponsor
Other Study IDs: BASEC 2019-01461
Record Dates: First submitted 2019-10-07; First posted 2019-10-11 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Sarcopenia
Keywords: Prevalence; Sarcopenia; Geriatric
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess the prevalence of sarcopenia among inpatients on acute geriatrics and geriatric rehabilitation wards of a Swiss university department of geriatric medicine using the most recent diagnosis definitions from european guidelines.

ELIGIBILITY:
Inclusion Criteria:

- All patients >65 years old admitted to acute geriatrics and geriatric rehabilitation at the study site

Exclusion Criteria:

* Lack of informed written consent
* Implanted defibrillation device
* Acute Sepsis, severe volume overload or dehydration
* Life expectancy of < 3 months according to treating physician
* Unremovable bandages
* Patients in isolation rooms on the ward
* Measurement is not possible due to organizational reasons
* Inability to follow the procedures, e.g. due to language problems, psychological disorders

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population will be selected by the University Department of Geriatric Medicine FELIX PLATTER
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Presence of Sarcopenia (yes/no) | Baseline
  Using EWGSOP2 cut-off points
Muscle quantity, measured by Body Impedance Analysis (kg) | Baseline
Hand Grip Strength (kPa) | Baseline
Gait Speed (m/s) | Baseline
Timed up and go Test (s) | Baseline

SECONDARY OUTCOMES:
Mini Mental Status (Score range from 0 to 30 Points; higher scores reflect better cognitive status) | Baseline
Nutritional risk Screening (Score range from 0 to 7 Points; higher scores reflect higher risk of malnutrition) | Baseline
Geriatric Depression Scale short version (Score range from 0 to 6 Points; higher scores reflect higher risk of depression) | Baseline
Functional Independence Measure at Admission (Score range from 18 to 126 Points; higher scores reflect better functionality) | Baseline
Calf and Mid-upper arm Circumference (cm) | Baseline
Body Mass Index (kg/m^2) | Baseline
  Weight and height will be combined to report Body Mass Index in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Dominic K. Bertschi, Dr., Principal Investigator — University Department of Geriatric Medicine FELIX PLATTER; Caroline Kiss, Dr., Study Chair — University Department of Geriatric Medicine FELIX PLATTER; Reto W. Kressig, Prof. Dr., Study Director — University Department of Geriatric Medicine FELIX PLATTER
Locations (1):
- University Department of Geriatric Medicine FELIX PLATTER, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No